CLINICAL TRIAL: NCT06550479
Title: Comparison of Tree Types of Distal Arteriovenous Fistulas: Snuffbox Fistula (SBAVF), Radiocephalic Fistula (RCAVF) and RCAVF With Venous Branch Patch.
Brief Title: Comparison of Three Types of Distal Arteriovenous Fistulas: SBAVF, RCAVF, and RCAVF With Venous Branch Patch.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WMU
Record Dates: First submitted 2024-07-30; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Dialysis; Complications; Vascular Access Complication

STUDY DESIGN:
Intervention Model Description: Comparison of three different distal AVF types
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SBAVF (Experimental): Patients enrolled for snuffbox fistula creation.
  Interventions: Procedure: AVF
- RCAVF (Experimental): Patients enrolled for RCAVF
  Interventions: Procedure: AVF
- RCAVF with venous branch patch (Experimental): Patients enrolled for RCAVF with venous branch patch
  Interventions: Procedure: AVF

INTERVENTIONS:
Procedure: AVF — Distal forearm AVF for hemodialysis.

SUMMARY:
This study aims to determine which type of distal arteriovenous fistula (SBAVF, RCAVF, and RCAVF with venous branch patch) is most clinically favorable.

The recommendations and scientific evidence do not suggest which option should be chosen initially.

The investigators expect that results will show which type of the anastomosis should be preferred.

DETAILED DESCRIPTION:
Research Project Objectives An important aspect in maintaining hemodialysis therapy is an optimal vascular access (AV) in patients with end-stage renal disease (ESRD). The radiocephalic arteriovenous (RCAVF), at the level of the wrist, or snuffbox fistula SBAVF stands out as the preferred vascular access (VA) for hemodialysis, due to its lower risk of infection and mortality compared to alternative options. The inherent properties of AVFs contributes not only to improved patient's safety but also to more efficient hemodialysis procedures. Despite this, AVFs has two disadvantages: a high early failure rate, occurring within one month after access creation, and a high failure rate during a maturation. Early failure rates differ between groups, ranging from 2-23% in brachiocephalic AVF (BCAVF) to up to 5-46%, in RCAVFs.[1] In the Jemcow study , a fistula was defined as mature when blood flow was greater than 500 ml/min and diameter of the cephalic vein exceeded 5 mm. Depending on when AVFs attained maturity, 53% of patients had successful AVF maturation, 36% had prolonged maturation i.e., within eight weeks, and 11% of AVFs failed to mature. Female sex, older patients, poor upper extremity vessels, distal placements and accesses with smaller diameter artery and vein are risk factors for failure to mature.

Despite advances in surgical techniques and perioperative care, fistula maturation remains a challenging part of hemodialysis access. This was shown by Bylsma et al., who conducted a meta-analysis that raised doubt on the AVF's utility in addressing ESRD.3 They evaluated the outcomes of more than 60.000 AVF access formations and found 1-year primary, primary assisted, and secondary patency rates of 64%, 73%, and 79%, respectively. However, only 26% of created fistulas were reported as mature at 6 months and 21% of fistulas were abandoned without use. In another meta-analysis study by Al-Jaishi, based on 37 studies, the risk of primary failure was 23% and primary patency rate was 60% at 1 year and 51% at 2 years.4 Clinical fistula maturation is the result of a crucial process in establishing functional VA for hemodialysis patients. It refers to the formation of a mature, useable AVF supplying the necessary blood volume for efficient dialysis. Data from a multicentre perspective cohort study by Robbin et al. of 602 patients who received a new single-stage AVF, demonstrated that unassisted and overall AVF clinical maturation can be predicted by three ultrasound parameters, fistula blood flow, diameter and depth. Performing such assessment, 6 weeks after surgery, provides valuable guidance regarding early intervention to facilitate maturation (e.g., percutaneous angioplasty or early planning of a second anastomosis) may increase maturation/utilization of the fistula and reduce exposure to central venous catheters.

The study will enroll individuals with and chronic kidney disease (CKD) in stage G4 and G5 including hemodialysis (HD) patients.

Clinical practice guidelines recommend distal arteriovenous fistula (AVF) RCAVF or SBAVF, rather than proximal arteriovenous anastomosis involving the brachial artery due to high risk of hemodialysis access hand ischemia and high flow heart failure. There have been no studies comparing the three aforementioned distal anastomosis in a single project.

Research hypothesis: There are differences between various types of AVF with regard to of early and late patency rates. The investigators also suppose that the type of AVFs may influence the postoperative increase in arteriovenous fistula diameter, blood flow, and, finally, AVF maturation.

Working second hypothesis: Demographical and clinical characteristic of the patients may have impact on AVF success rate and maturation.

Secondary objective of this study is to perform enhanced assessments of arterial health preoperatively and correlate these measurements with vascular lesions.

Work plan Participants will be subjects of a thorough evaluation of the morphological state of upper limb vessels by the techniques presented in the methodology of the study. The study plan foresees the recruitment of patients, whose will have their vessels of the upper limbs carried out in-depth assessment. Then creation of the vascular access - arteriovenous fistula for dialysis, will be performed. The choice of arteriovenous fistula type (SBAVF, RCAVF, and RCAVF with venous branch patch) will depend on the vascular anatomy obtained by Doppler ultrasonography.

AVF maturation will be evaluated after 6 weeks post-surgery using Doppller ultrasound. A fistula was considered mature when the blood flow exceeded 500 ml/min and the diameter of the cephalic vein exceeded 5 mm.

Study design Prospective study with recruitment of consecutive approximately 3 x 60 patients with chronic kidney disease stage 4 or 5, who will be referred for vascular access creation for hemodialysis.

Inclusion: (1) Aged >18 years, (2) has chronic kidney disease with estimated glomerular filtration rate (eGFR) <20 mL/min/1.73 m2 , (3) is undergoing AVF creation with venous end-to-arterial side anastomosis in the upper extremity.

Exclusion: (1) Heart failure of New York Heart Association functional class III or IV, and (2) episode of cardio- or cerebrovascular event or receiving intervention therapy within 3 months prior to screening. (3) had the primary anastomosis in the past on ipsilateral extremity After obtaining an informed consent to participate in the study each participant will be tested with followed measures.

Study measures Demographic and clinical characteristic will be collected during interview (family longevity, hospitalizations, history of vein cannulation) and based on medical records (cardiac events including angiographic studies, cancer, diabetes, peripheral artery diseases, dementia and other co-morbidities). Physical examination focused on heart function (blood pressure in two positions, heart rate, congestion in auscultation and chest as well as vascular anatomy examination with Allen test (patency of palmar arch), pulse presence, veins patency with and without stasis.

Imaging studies Ultrasound condition of vessel will be evaluated prior AVF creation (upper arms flow, diameter of arteries and veins, possible stenosis, etc) and in follow up period (day -1, 1 and 6 weeks). In selected cases (history of previous subclavian vein catheterization, collateral circulation developed) venography will be performed.

Whole blood parameters.

Blood samples will be taken at routine control, or before routine dialysis session in HD patients (referred for AVF placement).

Routine laboratory parameters collected at baseline and during follow-up (14-28, 56-60, 90 day): Complete blood counts with focus on neutrophil-lymphocyte ratio (NLR), phosphorus, calcium, parathormone, C-reactive protein (CRP), urea acid, lipids (cholesterol fractions, triglycerides).

Statistical analysis All participants data from recruitment and follow up will be collected in special designed computer program. The primary outcome of this study is AVF success (patent and mature) at 6 weeks post creation. Baseline patient characteristics including age, gender and co-morbidities will be compared between the patients with successful AVF and those with unsuccessful AVF. Categorical variables will be presented by frequency (percentage) and comparisons will be made via the Chi-square or Fisher's Exact test. Underlying distributions of continuous variables will be tested for normality using the Shapiro-Wilk test and then analyzed with appropriate tests. Kaplan-Meier analysis will be performed for primary, secondary and functional patency rate. All analyses will be performed by external statistical laboratory with high references. The professional statistical expertise is planned (PREST laboratory at Mathematical Institute in Wroclaw) with utilization of R package and Statistica 13 software.

ELIGIBILITY:
Inclusion Criteria:

* Aged >18 years
* Chronic kidney disease with estimated glomerular filtration rate (eGFR) <20 mL/min/1.73 m2

Exclusion Criteria:

* Heart failure of New York Heart Association functional class III or IV,
* Episode of cardio- or cerebrovascular event or receiving intervention therapy within 3 months prior to screening.
* The patient had the primary anastomosis in the past on ipsilateral extremity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Primary patency: | 12 months
  The interval between VA creation and the first re-intervention (intervention free VA survival) for VA dysfunction or thrombosis, the time of measurement of patency or the time of its abandonment
Assisted primary patency: | 36 months
  The interval between VA creation and the first occlusion (thrombosis free VA survival) or measurement of patency including operative/endovascular interventions to maintain the VA.
Secondary patency | 36 months
  The interval between VA creation and the abandonment of this VA (i.e. thrombosis) after one or more interventions or the time of measurement of patency including achievement of a censored event (death, change of HD modality, loss of follow-up).

SECONDARY OUTCOMES:
Mature VA | 6 weeks
  A fistula was considered mature when the blood flow exceeded 500 ml/min and the diameter of the cephalic vein exceeded 5 mm.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nephrology and Transplantation Medicine, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tordoir J, Canaud B, Haage P, Konner K, Basci A, Fouque D, Kooman J, Martin-Malo A, Pedrini L, Pizzarelli F, Tattersall J, Vennegoor M, Wanner C, ter Wee P, Vanholder R. EBPG on Vascular Access. Nephrol Dial Transplant. 2007 May;22 Suppl 2:ii88-117. doi: 10.1093/ndt/gfm021. No abstract available. PMID 17507428
- [Result] Roy-Chaudhury P, Kelly BS, Melhem M, Zhang J, Li J, Desai P, Munda R, Heffelfinger SC. Vascular access in hemodialysis: issues, management, and emerging concepts. Cardiol Clin. 2005 Aug;23(3):249-73. doi: 10.1016/j.ccl.2005.04.004. PMID 16084276
- [Result] Stoner L, Sabatier MJ. Use of ultrasound for non-invasive assessment of flow-mediated dilation. J Atheroscler Thromb. 2012;19(5):407-21. doi: 10.5551/jat.11395. Epub 2012 Mar 1. PMID 22659525
- [Result] Jemcov TK. Morphologic and functional vessels characteristics assessed by ultrasonography for prediction of radiocephalic fistula maturation. J Vasc Access. 2013 Oct-Dec;14(4):356-63. doi: 10.5301/jva.5000163. Epub 2013 Jul 1. PMID 23817950
- [Result] Bylsma LC, Gage SM, Reichert H, Dahl SLM, Lawson JH. Arteriovenous Fistulae for Haemodialysis: A Systematic Review and Meta-analysis of Efficacy and Safety Outcomes. Eur J Vasc Endovasc Surg. 2017 Oct;54(4):513-522. doi: 10.1016/j.ejvs.2017.06.024. Epub 2017 Aug 23. PMID 28843984
- [Result] Al-Jaishi AA, Oliver MJ, Thomas SM, Lok CE, Zhang JC, Garg AX, Kosa SD, Quinn RR, Moist LM. Patency rates of the arteriovenous fistula for hemodialysis: a systematic review and meta-analysis. Am J Kidney Dis. 2014 Mar;63(3):464-78. doi: 10.1053/j.ajkd.2013.08.023. Epub 2013 Oct 30. PMID 24183112